CLINICAL TRIAL: NCT00404482
Title: Efficacy and Adverse Effects of Cyclosporine A in the Treatment of Chronic Anterior Uveitis in Patients With Juvenile Idiopathic Arthritis
Brief Title: Cyclosporine A in the Treatment of Juvenile Idiopathic Arthritis (JIA) Associated Chronic Anterior Uveitis
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Other Study IDs: 01-1106
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Uveitis; Juvenile Idiopathic Arthritis
Keywords: uveitis; jia; Cyclosporine A; MTX
MeSH Terms: conditions — Uveitis; Arthritis, Juvenile | interventions — Cyclosporine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Cyclosporine A

SUMMARY:
Juvenile idiopathic arthritis (JIA) is often associated with chronic anterior uveitis. Presence of vision threatening complications may indicate immunosuppressive therapy. In this study, the experience with cyclosporine A (CsA) as mono- or combination-therapy is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* uveitis
* JIA

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with JIA and cyclosporin A therapy
Sampling Method: Probability Sample
Enrollment: 60
Dates: Start 1991-01; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Tappeiner, MD, Principal Investigator — Department of Ophthalmology at University Bern - Inselspital
Locations (3):
- Germany (3):
  - Deutsches Zentrum für Kinder- und Jugendrheumatologie, Garmisch-Partenkirchen
  - Department of Ophthalmology at St.-FranziskusHospital, Münster
  - Kinder und Jugendrheumatologie St. Josef Stift, Sendenhorst